CLINICAL TRIAL: NCT03072368
Title: Iris Colors in Neonates: Do They Really Change? Prevalence, Predicting Factors and Associated Characteristics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HYMC-0081-16
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Eye Color
MeSH Terms: interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blue eyes (Active Comparator): 50 babies born with blue eyes will be photographed and followed-up at baseline; 3 months and 12 months of age
  Interventions: Other: Photograph
- Brown eyes (Active Comparator): 50 babies born with brown eyes will be photographed and followed-up at baseline; 3 months and 12 months of age
  Interventions: Other: Photograph
- Green eyes (Active Comparator): 50 babies born with green eyes will be photographed and followed-up at baseline; 3 months and 12 months of age
  Interventions: Other: Photograph
- Hazel eyes (Active Comparator): 50 babies born with hazel eyes will be photographed and followed-up at baseline; 3 months and 12 months of age
  Interventions: Other: Photograph

INTERVENTIONS:
Other: Photograph — Babies will be photographed and eye color will be observed and documented at birth, 3 months and one year of age

SUMMARY:
The goal of our study is to examine eye color at birth and the longitudinal change in eye color of preterm and full-term newborns.

ELIGIBILITY:
Inclusion Criteria:

* Any baby born between the 24-42 week of gestation admitted to the well-baby nursery or the NICU whose parents have signed an informed consent.

Exclusion Criteria:

* Neonatal conjunctivitis
* Neonatal sepsis
* Inborn error of metabolism or genetic syndrome
* Eye abnormalities
* Parental refusal

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in eye color | One year
  Change will be measured according to a validated classification of blue/hazel/green or brown

CONTACTS AND LOCATIONS:
Overall Officials: Amit Hochberg, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No